CLINICAL TRIAL: NCT05850130
Title: A Multicenter, 2-cohort Phase II GERCOR Study to Evaluate the Interest of Acupuncture on Oxaliplatin-induced Peripheral Neuropathy in Patients With Gastro-intestinal Solid Tumors Who Discontinued Oxaliplatin-based Chemotherapy (ACUPOX)
Brief Title: Acupuncture for Oxaliplatin-induced Peripheral Neuropathy in Gastro-intestinal Cancer Patients
Acronym: ACUPOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACUPOX G-114
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Liver Cancer; Gastric Cancer; Pancreas Cancer; Esophagus Cancer
Keywords: acupuncture
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: A multicenter, 2-cohort phase II study:
  Cohort 1: randomization into Arm A = Experimental or Arm B = Control
  Cohort 2: a single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): 6 weeks of acupuncture once a week. At week 7, patients will be assessed for the primary endpoint Then ,the patient may receive an optional 6 weeks of acupuncture. This option of acupuncture continuation will be left to the patient choice in agreement with a physician acupuncturist.
  Interventions: Other: Acupuncture intervention
- Arm B (Active Comparator): 6 weeks without acupuncture. At week 7, patients will be assessed for the primary endpoint.
  Then, the patient will receive or not acupuncture intervention:
  * A mandatory acupuncture once a week if the patient' NRS global score at week 7 is ≥ 4 .
  * No acupuncture if the patient' NRS global score at week 7 is <4,
  Interventions: Other: No acupuncture

INTERVENTIONS:
Other: Acupuncture intervention — 6 weeks of acupuncture once a week. The acupuncture intervention will consist of weekly session administered over a period of 6 weeks (± 4 days). A two-way verum acupuncture treatment protocol will employ 8 selected acupoints.
  After week 7, patients included in Arm A may receive an optional 6 weeks of acupuncture. This option of acupuncture continuation will be left to the patient choice in agreement with a physician acupuncturist.
  Arms: Arm A
Other: No acupuncture — The patient in the Arm B will not receive acupuncture treatment for a period of 6 weeks after randomization (weeks 1-6) and during the following weeks 8-13 (acupuncture intervention) if its NRS score is <4/10 at week 7. If the patient' NRS score is ≥ 4/10 at week 7, the patient in control Arm B will receive the same acupuncture intervention that the patient in the Arm A (6 weeks).
  Arms: Arm B

SUMMARY:
ACUPOX is a multicenter, open label, 2-cohort based phase II clinical study evaluating the interest of a standardized protocol of verum acupuncture in treatment of Oxaliplatin-induced peripheral neuropathy in patients with gastro-intestinal solid tumors who discontinued oxaliplatin-containing chemotherapy.

DETAILED DESCRIPTION:
In this design, patients will be randomized into two-arm (2:1 allocation) Cohort 1: a comparative randomized design (Arm A = Experimental vs Arm B = Control) or included into Cohort 2: a single arm design.

The study follows the Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA) guideline.

All acupuncture interventions will be conducted by a physician acupuncturist. If the patient will be getting chemotherapy (that is optional treatment) during the study duration, acupuncture will be given at the same time.

ELIGIBILITY:
Inclusion Criteria

Patient is included if:

1. Agree to participate in this study, voluntarily signing a written informed consent form,
2. Aged ≥ 18 years,
3. Have an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2,
4. Have histologically or cytologically confirmed gastro-intestinal solid tumors, previously treated with any oxaliplatin-based chemotherapy; a concomitant radio-chemotherapy course is allowed,
5. Had the last oxaliplatin infusion > 2 weeks before inclusion,
6. Present OIPN with a numerical rating score (NRS) ≥ 4/10 at inclusion,
7. Currently receiving or recently completed chemotherapy (adjuvant, neoadjuvant, or advanced stage). Patients may receive current chemotherapy treatment (e.g., with FOLFIRI, 5-fluorouracil, bevacizumab regimens), excluding platinum salts and taxane-based regimens during the study,
8. Are able to understand/read French,
9. Are registered in a national health care system (PUMa - Protection Universelle Maladie included),

Exclusion Criteria

Patients is excluded if:

1. Had acupuncture sessions for the prevention of chemotherapy-induced side effects in the last 3 months prior to inclusion,
2. Had previous and/or current chemotherapy treatments with taxane-based regimens (e.g., the TFOX regimen [docetaxel, oxaliplatin, leucovorin, and 5-fluorouracil]),
3. Have a history of preexisting clinically-significant peripheral neuropathy due to any cause other than chemotherapy (borrelia infection, human immunodeficiency virus infection, hereditary factors, tumor compression, nutritional deprivation, alcohol, diabetes, etc.),
4. Have a recent history (within 4 weeks prior to start of acupuncture) of abusing alcohol, prescription, or illicit drugs (including cannabinoid), or medical, psychological, or social conditions that may interfere with the patient's compliance with the study intervention, NB: The patient should be informed that drinking alcohol should be avoided while on study.
5. Have any other condition that, in the opinion of the investigator, is unstable or could jeopardize the safety of the patient and her/his compliance during the study,
6. Have limb edema of grade 3 (CTCAE v5),
7. Had phytotherapy within 2 weeks before a week 1-14 intervention,
8. Are pregnant or breastfeeding,
9. Are under the tutorship or guardianship of the state or in custody of the justice system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-point improvement in the global NRS | Week 7
  The primary endpoint is a 2-point improvement in the global numeric rating scale (NRS) score from randomization/inclusion defined by the patient at week 7. The 11-point NRS range from 0 to 10 (0 = no symptom, 1-3 = mild, 4-6 = moderate, 7-10 = severe).

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) score | Week 7
  A success of acupuncture for the patient is defined by a 2-point improvement on the overall NRS between baseline and week 7 after the randomization of Cohort 1 and inclusion of Cohort 2.
Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy twenty-item scale (QLQ-CIPN20) questionnaire | Assess at baseline, at week 7, 14, and at 6 months
  The EORTC QLQ-CIPN20 questionnaire consists of 20 items that are divided into 3 subscales: the items in CIPN20 have been divided into three subscales. The sensory subscale consists of items 1, 2, 3, 4, 5, 6, 9, 10, and 18; motor: items 7, 8, 11, 12, 13, 14, 15, and 19; and autonomic nerve-related: items 16, 17, and 20. Each subscale is summed and linearly transformed to a score that can range from 0 to 100, where higher scores represent greater CIPN symptom severity. Patients will rate their experience for each symptom during the previous week using scores from 1 (not at all) to 4 (very much).
Brief Pain Inventory (BPI) score | Assess at baseline, at week 7, 14, and at 6 months
  This 9-item BPI self-reported questionnaire provides information on the intensity of pain and the degree to which pain interferes with function. Pain is rated over the prior week and the degree to which the pain interferes with activities using a 0 to 10-point scale.
Peripheral sensory neuropathy grading scale | Assess at baseline, at each intervention visit, at week 7, 14, and at 6 months
  Severity of the peripheral sensory neuropathies will be classified using a 4-point scale ranging from grade 1 to grade 4 per criteria established in NCI CTCAE v. 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Kempf, MD, Principal Investigator — Henri Mondor University Hospital
Locations (5):
- France (5):
  - Centre intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Institu Daniel Hollard, Grenoble
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris